CLINICAL TRIAL: NCT05173428
Title: The Effect of Online Motivational Interviews Based on the Transtheoretical Model on Pregnant Women's Prediction of Smoking Cessation Success, Self-Efficacy Levels and Smoking Cessation Behaviors
Brief Title: The Effect of Motivational Interviews Based on the Transtheoretic Model on Pregnant Women's Smoking Cessation Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Betul Esra Cevik, Research Assistant, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SCU-BECEVIK-001
Record Dates: First submitted 2021-12-09; First posted 2021-12-30 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Smoking Cessation; Smoking, Tobacco
Keywords: Motivational Interviews; Transtheoretic Model; Pregnancy
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In a randomized controlled study, blinding will be done in terms of statistician and reporting. Research data will be encoded and transferred to the computer without specifying the intervention and control group (for example; A group and B group). The analysis of these data coded in terms of groups will be done by a statistician. After the statistical analysis is done and the research report is written, the researcher will explain the coding for the intervention and control group. In this way, detection bias, statistical bias and reporting bias will be controlled.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Gruop (Experimental): Online motivational interviews based on the transtheoretic model with the intervention group will be held via zoom. Data collection forms will be applied to the intervention group at the first interview, at the 3rd month as an interim monitoring, and at the 6th month as the final monitoring.
  Interventions: Behavioral: Smoking Cessation Program Based on Transtheoretic Model
- Control Gruop (No Intervention): No intervention will be made to the control group, and data collection forms will be applied at the first interview and 6 months after the first interview.

INTERVENTIONS:
Behavioral: Smoking Cessation Program Based on Transtheoretic Model — Conducting motivational interviews based on the transtheoretic model according to the stages of change that individuals are in.
  Arms: Interventional Gruop

SUMMARY:
This study is planned to determine the effect of online motivational interviews based on the transtheoretic model on the prediction of smoking cessation success, self-efficacy levels and smoking cessation behavior of pregnant women.It is an experimental research.

DETAILED DESCRIPTION:
The population of the research will be the pregnant women registered in the family health center in Sivas city center.The sample of the study will consist of pregnant women who smoke and agree to participate in the study.Power analysis was calculated using G * Power 3.1.9.2 program. With 76% effect size, 90% power and 0.05 significance level, the required sample size was determined as 30 individuals per group, and 60 individuals in total. It was decided to include 66 individuals, 33 individuals in the intervention group and 33 individuals in the control group, by taking 10% more of the calculated sample against the possibility of sample loss during the study.Smoking Cessation Success Prediction Scale Self-Efficacy Level Scale Decision-Making Balance Scale Behavior Change Stage Diagnostic Questionnaire Fagerström Nicotine Addiction Test will be used as measurement tools.Pregnant women who agree to participate in the study will fill in the Informed Consent Form and other measurement tools.Interviews with the pregnant women in the intervention group will be held face-to-face via the Zoom application for a total of 6 times.Data collection forms will be applied to the control group at the first interview and at the last interview (6 months later), and for the intervention group at the first interview, 3 months and 6 months later, a total of 3 times.After each assessment moment, the data obtained will be exported to the "Statistical Package for Social Sciences Software" (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Not completing the 16th week of pregnancy
* Being 18 years or older
* To smoke at least 1 cigarette a day
* Being able to use a smart phone or computer and having internet
* Being literate

Exclusion Criteria:

* Unable to use a computer or smartphone
* Being at the 17th and above gestational week
* Having any mental illness
* Illiterate pregnant women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Smoking-Cessation Success Prediction Scale | 6 months
  The scale consists of 10 items.Items in the scale are evaluated with a 5-point Likert scale (1: too little, 2: little, 3: middle, 4: a little too much, 5: much).The maximum score that can be obtained from the scale is 50, and the minimum score is 10. Scale score indicates that the success of smoking cessation will be high.
Decisional Balance Scale | 6 months
  The scale, which has 24 items, consists of two sub-dimensions: "Positive aspects of smoking" and "Negative aspects of smoking". Each item of the scale is scored from 1 to 5 as 1- I strongly disagree, 2- I do not agree, 3- I neither agree nor disagree, 4- I agree, 5- I completely agree.For both sub-dimensions, the minimum score that can be obtained from the scale is 12, and the maximum score is 60.Scale total score; It is calculated by subtracting the perceived harm total score of smoking from the total perceived benefit score of smoking. The negative (-) result indicates that the perceived harms of smoking are dominant in the decision-making balance. The positive (+) result indicates that the perceived benefits of smoking are dominant in the decision-making balance.
Self-Efficacy Level Scale | 6 months
  The scale consists of 23 items and 4 sub-dimensions: starting the behavior, maintaining the behavior, completing the behavior and struggling with obstacles.For each item in the scale; 1-Does not describe me at all, 2-Describes me a little, 3-I am undecided, 4-Describes me well, 5-Describes me very well.A minimum of 23 and a maximum of 115 points can be obtained from the scale. The high total score obtained from the scale indicates that the general self-efficacy perception is high.
Fagerstrom Test For Nicotine Dependence | 6 months
  The test was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence.
  In scoring the Fagerstrom Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.

CONTACTS AND LOCATIONS:
Overall Officials: Semra ZORLU, PhD, Study Director — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)